CLINICAL TRIAL: NCT00131833
Title: Typhoid Vi Vaccine Effectiveness in a Population Older Than 5 Years of Age Living in an Endemic Area in Hechi, Guangxi, P.R. China: A Group-Randomized Controlled Demonstration Project
Brief Title: Typhoid Vi Vaccine Effectiveness in Hechi, Guangxi, China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Hechi City Center for Disease Centrol (Unknown); Wellcome Trust (Other); University of Western Ontario, Canada (Other)
Responsible Party: Mr. Leon Ochiai, International Vaccine Institute
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: T3
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Typhoid; Paratyphoid Fever
Keywords: salmonella; typhoid vaccine; enteric fever
MeSH Terms: conditions — Typhoid Fever; Paratyphoid Fever | interventions — Vi polysaccharide vaccine, typhoid

INTERVENTIONS:
Biological: Typhoid Vi vaccine
Biological: Meningococcal A (control)

SUMMARY:
This study is part of International Vaccine Institute (IVI)'s typhoid Vi demonstration project that aims to accelerate the rational introduction of Vi vaccines in typhoid endemic countries. The purpose of this study is to determine the effectiveness of the Vi vaccine following a mass typhoid immunization campaign in an endemic area in Hechi City in the Guangxhi province of China. The cost-effectiveness and safety of Vi vaccination will also be evaluated.

DETAILED DESCRIPTION:
Typhoid fever is a major cause of morbidity worldwide. The disease predominantly affects school-aged children, is more prevalent in urban areas, may last for several weeks and can lead to serious complications. Management of this disease is further complicated by the emergence of multi-drug resistant strains. Vaccination of high risk populations is considered the most promising strategy for the control of typhoid fever. The Vi polysaccharide vaccine has been targeted for accelerated introduction into public health programs due to the following reasons: it has been shown to have consistent efficacy results even in areas of high typhoid incidence, is given as a single dose, lacks patent protection and requires less strict cold chain requirements.

This project attempts to evaluate a new vaccination strategy for residents of endemic areas. A cluster-randomized trial involving the Vi polysaccharide vaccine and an active control (meningococcal A vaccine) was designed to determine the effectiveness and the feasibility of providing Vi vaccine under actual programmatic conditions in 2 populous townships of Hechi City. The vaccines used in this study are locally produced and licensed in China. A 1 year pilot phase will precede the actual Vi-demonstration project. Surveillance for typhoid fever cases will continue after the mass immunization campaign. A passive surveillance system to evaluate adverse events following immunization will be implemented. Socio-economic studies will be conducted in parallel to the effectiveness evaluation. The knowledge, attitudes, beliefs and practices among parents and health care providers regarding typhoid illness, treatment and prevention will be assessed. Logistic, feasibility and vaccine costs will also be determined.

Secondary objectives of this trial are:

* To estimate the logistic feasibility of a mass typhoid immunization campaign
* To assess the knowledge, attitudes, beliefs and practices among parents and health care providers regarding typhoid illness, treatment and prevention
* To study typhoid fever risk factors in the population

ELIGIBILITY:
Inclusion Criteria:

* Registered in the project census

Exclusion Criteria:

* Pregnant
* Lactating
* Fever > 37.5 degrees Celsius, axillary

Ages: 5 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 96468
Dates: Start 2001-10; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
vaccine effectiveness
cost effectiveness of typhoid Vi immunization
adverse events

SECONDARY OUTCOMES:
logistic feasibility of mass typhoid immunization
anti-Vi antibody response
knowledge, attitudes, beliefs and practices of parents and health care providers on typhoid fever prevention and treatment
Typhoid risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Dong Baiqing, MD, Principal Investigator — Guangxi Center for Disease Control and Prevention
Locations (1):
- Hechi City Center for Disease Control, Hechi, Guangxi, China

REFERENCES:
- [Background] Dong BQ, Yang J, Tang ZZ, Yang HH, Zeng J, Zhang J, Wang ML, Liang GC, Si GA, Li CY, Liang DB, Liao HZ, Ochiai RL, Mohammad A, Acosta CJ, Clemens J. [Application of cluster randomization method on typhoid Vi vaccine trails]. Zhonghua Liu Xing Bing Xue Za Zhi. 2005 Feb;26(2):97-100. Chinese. PMID 15921608
- [Background] Yang J, Acosta CJ, Si GA, Zeng J, Li CY, Liang DB, Ochiai RL, Page AL, Danovaro-Holliday MC, Zhang J, Zhou BD, Liao HZ, Wang ML, Tan DM, Tang ZZ, Gong J, Park JK, Ali M, Ivanoff B, Liang GC, Yang HH, Pang T, Xu ZY, Donner A, Galindo CM, Dong BQ, Clemens JD. A mass vaccination campaign targeting adults and children to prevent typhoid fever in Hechi; expanding the use of Vi polysaccharide vaccine in southeast China: a cluster-randomized trial. BMC Public Health. 2005 May 18;5:49. doi: 10.1186/1471-2458-5-49. PMID 15904514
- [Background] Acosta CJ, Galindo CM, Ochiai RL, Danovaro-Holliday MC, Page AL, Thiem VD, Park JK, Park E, Koo H, Wang XY, Abu-Elyazeed R, Ali M, Albert MJ, Ivanoff B, Pang T, Xu ZY, Clemens JD. The role of epidemiology in the introduction of vi polysaccharide typhoid fever vaccines in Asia. J Health Popul Nutr. 2004 Sep;22(3):240-5. PMID 15609776